CLINICAL TRIAL: NCT07208344
Title: A Randomized Double-blind Clinical Study on the Use of Umbilical Cord Blood as an Adjuvant Therapy to Improve Cognitive Function in Alzheimer's Disease and Its Mechanism of Action
Brief Title: Intravenous Infusion of Umbilical Cord Blood as an Adjunctive Treatment for Alzheimer's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Collaborators: Shandong Qilu Stem Cell Engineering Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHSL-QLGXB-MNC-AD
Record Dates: First submitted 2025-09-02; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease (AD)
MeSH Terms: conditions — Alzheimer Disease | interventions — Rivastigmine; Galantamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): The conventional treatment plan was supplemented with intravenous injection of normal saline (in a blinded manner)
  Interventions: Drug: Conventional medical treatment：donepezil, rivastigmine or galantamine
- Low-dose group (Experimental): In addition to the conventional treatment regimen, intravenous infusion of umbilical cord blood mononuclear cells (1×10^8 cells per infusion) will be administered. The infusions will be carried out via the intravenous route at one - week intervals for a total of four consecutive times. One month after the completion of the fourth infusion, the fifth infusion will be performed.
  Interventions: Biological: Intravenous infusion of mononuclear cells from umbilical cord blood; Drug: Conventional medical treatment：donepezil, rivastigmine or galantamine
- High-dose group (Experimental): In addition to the conventional treatment regimen, intravenous infusion of umbilical cord blood mononuclear cells (3×10^8 cells per infusion) will be administered. The infusions will be carried out via the intravenous route at one - week intervals for a total of four consecutive times. One month after the completion of the fourth infusion, the fifth infusion will be performed.
  Interventions: Biological: Intravenous infusion of mononuclear cells from umbilical cord blood; Drug: Conventional medical treatment：donepezil, rivastigmine or galantamine

INTERVENTIONS:
Biological: Intravenous infusion of mononuclear cells from umbilical cord blood — When performing cell infusion, it is essential to use an infusion set and follow the standard blood transfusion procedures. Before, during, and after the infusion, monitor the patient's body temperature, pulse, breathing, and blood pressure. When infusing cells, first flush the tube with 20-30 ml of 0.9% sodium chloride, and start the infusion at a rate of 20-30 drops per minute. After half an hour, if there are no adverse reactions, increase the rate to 30-50 drops per minute. During the cell infusion process, gently shake the cell bag once every 15 minutes. After the infusion is completed, flush the cell preservation bag with 20 ml of 0.9% sodium chloride and gently shake it. After that, use 0.9% sodium chloride to rinse the infusion set to remove the cells completely, to ensure the quantity of cell infusion.
  Arms: High-dose group; Low-dose group
Drug: Conventional medical treatment：donepezil, rivastigmine or galantamine — The treatment is carried out using drugs such as cholinesterase inhibitors (ChEI) which are suitable for mild to moderate Alzheimer's disease. For example, donepezil, rivastigmine, galantamine, etc. The frequency and dosage of drug administration should be in accordance with the instructions provided by the drug manufacturer.The patient should maintain the stability of the medication regimen throughout the entire study period.

SUMMARY:
This study is a single-center, prospective, double-blind, randomized controlled clinical trial (RCT).

Employing a parallel-group design, the trial plans to enroll 30 clinically diagnosed AD patients, who will be randomly assigned via a computerized randomization tool into three equal groups: low-dose, high-dose, and control (10 patients per group).

The blinded clinical trial consists of three phases:

**Screening Phase**: All enrolled patients must provide fully informed consent and meet inclusion criteria while avoiding exclusion criteria. Baseline assessments will be recorded, and single-cell omics samples will be collected. Patients may voluntarily opt for cerebrospinal fluid (CSF) sampling.

The umbilical cord blood (UCB) used clinically is sourced from the Shandong Cord Blood Hematopoietic Stem Cell Bank. Following erythrocyte and granulocyte depletion via lymphocyte separation and density gradient centrifugation, the UCB is purified to reduce immunogenicity and undergoes genetic screening to exclude the APOE4 risk allele.

**Treatment Phase**: In addition to standard care, patients will receive intravenous infusions at weekly intervals for four sessions. A fifth infusion will be administered one month after the fourth. The low-dose group receives 1×10⁸ UCB-derived mononuclear cells (UCB-MNCs) per infusion, the high-dose group receives 3×10⁸ UCB-MNCs, and the control group receives an equivalent volume of saline placebo.

All clinically administered UCB-MNCs undergo genetic screening to exclude the APOE4 risk allele.

**Follow-up Phase**:

Assessments will be conducted at 30 days (1 month), 60 days (2 months), 90 days (3 months), and 180 days (6 months) post-initial infusion, including:

1. CDR-SB scale scoring;
2. Total and subdomain scores of the Activities of Daily Living (ADL) scale;
3. Serum inflammatory cytokines (IL-1, IL-2, IL-6, IL-8, IL-10, TNF-α), AD biomarkers (P-tau181, P-tau217), and other relevant markers;
4. Single-cell omics sample collection;
5. Optional CSF sampling per patient preference.

After database lock, unblinding will occur for subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 50 - 75 years old, gender not restricted;
* Patients diagnosed with Alzheimer's disease (AD) according to the AT(N) diagnostic framework (with positive amyloid protein PET test results);
* MMSE score between 15 and 30 points, patients with mild to moderate Alzheimer's disease;
* The patient has a fixed caregiver who is willing to accompany the patient throughout the corresponding program;
* The patient has a literacy level above primary school, sufficient to complete the tests stipulated in the program;
* The patient or the guardian consents to participate in this clinical trial voluntarily and signs the informed consent form.

Exclusion Criteria:

* Dementia caused by other diseases, such as vascular dementia, frontotemporal dementia, and Lewy body dementia, etc.;
* The patient has other major systemic diseases, malignant tumors, chronic obstructive pulmonary disease or pulmonary fibrosis, etc. related to the lungs;
* The patient's white blood cell and neutrophil levels are below the normal lower limit;
* The patient has active infectious diseases, such as syphilis, AIDS, hepatitis B, hepatitis C;
* The patient has a history of stroke, epilepsy, alcohol abuse, or abuse of psychotropic drugs;
* Severe visual or hearing impairment, or those who cannot complete the relevant assessment due to other reasons;
* Patients who have participated in other clinical trials within the last 2 months;
* Other situations that the researchers consider not suitable for participating in clinical research.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) | Baseline, 1st, 2nd, 3rd and 6th month after treatment
  The Clinical Dementia Rating Scale-Sum of Boxes (CDR-SB) assesses cognitive functions through six different sub-items, including memory, orientation, judgment and problem-solving ability, social skills, family life and hobbies, and self-care ability.
  The total score of CDR-SB ranges from 0 to 18. The higher the score, the worse the patient's cognitive function and daily living ability.
  This helps to provide a more comprehensive understanding of the patient's cognitive functions in all aspects.
  The assessors need to undergo professional training, be familiar with the assessment methods and scoring criteria, and avoid being influenced by subjective factors in the assessment results.
  During the assessment process, it is necessary to have adequate communication with the respondents and caregivers to understand the medical history and living conditions, in order to obtain more accurate information.
Activity of Daily Living Scale（ADL） | Baseline, 1st, 2nd, 3rd and 6th month after treatment
  Activity of Daily Living Scale（ADL） is commonly used to assess the daily living abilities of the elderly, and it plays a crucial role in the screening of Alzheimer's disease (AD) and mild cognitive impairment (MCI).
  The minimum score is 16 (which is completely normal). Scores above 16 indicate varying degrees of functional decline, with the maximum being 56.
  The ADL scale consists of 14 items and is divided into two parts: the first part is the self-care scale for physical activities, including activities such as using the toilet, eating, dressing, daily hygiene, walking, and bathing. The second part is the instrumental daily living ability scale, including activities such as making phone calls, shopping, cooking, housework, taking public transportation, taking medicine, and managing finances.

SECONDARY OUTCOMES:
Serum levels of AD markers (P-tau181, 217) | Baseline, 1st, 2nd, 3rd and 6th month after treatment
  The level of P-tau 181 shows a strong correlation with the density of Tau tangles in the brain. The levels of P-tau 181 in the cerebrospinal fluid and blood of patients with Alzheimer's disease were significantly higher than those of patients with other neurodegenerative diseases and the normal population. The increase in P-tau 217 is closely related to another core pathological feature of the brain - the deposition of β-amyloid plaques.
  At the corresponding time point, blood samples (1.5 - 3 mL) were taken from the patients, and the levels of P-tau 181 and P-tau 217 were quantified using chemiluminescent enzyme immunoassay (cLEIA).
Cerebrospinal fluid(CSF) levels of AD markers (P-tau181, 217) | Baseline, 2nd month after treatment
  The level of P-tau 181 shows a strong correlation with the density of Tau tangles in the brain. The levels of P-tau 181 in the cerebrospinal fluid and blood of patients with Alzheimer's disease were significantly higher than those of patients with other neurodegenerative diseases and the normal population. The increase in P-tau 217 is closely related to another core pathological feature of the brain - the deposition of β-amyloid plaques. At the corresponding time point, a sample of the patient's cerebrospinal fluid (1-2 mL) was collected, and the levels of P-tau 181 and P-tau 217 in it were quantified using chemiluminescent enzyme immunoassay (cLEIA).
Minimum Mental State Examination（MMSE）Scores | Baseline, 1st, 2nd, 3rd and 6th month after treatment
  MMSE, which stands for Mini-Mental State Examination, was developed by Forstmann et al. in 1975 and is a widely used cognitive function screening tool in clinical and research settings. Its main purpose is to quickly and effectively assess the cognitive status of the subjects, especially to screen for the presence of cognitive impairments (such as dementia).
  The lowest score on the scale is 0 (indicating the most severe condition), and the highest score is 30 (indicating complete normality).
Montreal Cognitive Assessment（MoCA） | Baseline, 1st, 2nd, 3rd and 6th month after treatment
  The Montreal Cognitive Assessment (MoCA) scale was developed by Professor Nasreddine in 2004 as an assessment tool for rapid screening of mild cognitive impairment (MCI). The cognitive domains evaluated include attention and concentration, executive function, memory, language, visuospatial skills, abstract thinking, calculation and orientation. The total score of the scale is 30 points, with the lowest score being 0. The higher the score, the better the performance of the test subject. The test result is considered normal if it is ≥ 26 points.
Alzheimer disease assessment scale-cognitive component (ADAS-Cog) | Baseline, 1st, 2nd, 3rd and 6th month after treatment
  The Alzheimer disease assessment scale - cognitive component (ADAS-cog) is one of the most widely used general cognitive measurement methods in clinical trials of Alzheimer's disease. It consists of 12 items and can assess the severity of cognitive symptoms in AD and changes in treatment. It is often used for the efficacy evaluation of mild to moderate AD (typically, a 4-point improvement is regarded as the clinical criterion for the effectiveness of the drug). The total score of this scale ranges from 0 (no errors or no damage) to 70 (severe damage).
tau-Positron Emission Tomography（tau-PET） | Baseline, 3rd and 6th month after treatment
  Tau-PET can specifically bind to abnormal tau proteins through intravenous injection, and directly visualize the distribution and density of neurofibrillary tangles (one of the core pathological features of Alzheimer's disease) in the brain in real time.Inspection process: A radioactive tracer is injected into the vein of the subject, and then the subject is left to wait for a period of time for the tracer to distribute in the brain. Finally, a PET scan is conducted to generate images.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of the University of Science and Technology of China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No